CLINICAL TRIAL: NCT05310227
Title: A Prospective, Single Arm, Open Label Study of the Safety and Efficacy of Nerivio™ for the Acute Treatment of New Daily Headache Persistence (NDHP) in Adolescents
Brief Title: Nerivio Device for Treatment of New Daily Headache Persistence (NDHP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The device became FDA approved during enrollment thereby nullifying the need to complete the trial. No clinical data was collected.
Sponsor: Children's National Research Institute (Other)
Collaborators: Theranica (Industry)
Responsible Party: Principal Investigator, Marc DiSabella, Principal Investigator, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016835
Record Dates: First submitted 2022-03-21; First posted 2022-04-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: New Daily Persistent Headache (NDPH)
Keywords: New Daily Persistent Headache (NDPH); Nerivio Device

STUDY DESIGN:
Intervention Model Description: The device is a wireless wearable battery-operated stimulation unit controlled by a dedicated smartphone application. Treatments with Nerivio™ are self-administered by the user at the onset of a headache. The Nerivio™ includes several main components:
  * A pair of electrodes covered with hydrogel and a removeable protective film
  * An electronic circuitry and a battery
  * A software that includes firmware and a software application for mobile platforms
  * An armband to secure the attachment of the device and enable a discreet treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Participants will receive a device and will be asked to treat headaches with it and report in the app the characteristics of the attacks at the beginning of the attack as well as at 2 hours after the treatment.
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — The device is a wireless wearable battery-operated stimulation unit controlled by a dedicated smartphone application. Treatments with Nerivio™ are self-administered by the user at the onset of a headache

SUMMARY:
The goal of this study is to examine the effects of the Remote Electrical Neuromodulation (REN) device on adolescents ages 12-17 who have been diagnosed with New Daily Persistent Headache (NDPH). Pediatric patients with a diagnosis of new daily persistent headache are typically resistant to standard pharmacologic treatments and often experience systemic side effects related to medications; thus, REN offers the potential for an exciting new treatment option for patients with refractory headache disorders. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. Ultimately, the investigators hope to gain insights into the safety and efficacy of Nerivio™ for the acute treatment of NDPH in adolescents. The goal of this study is to demonstrate headache relief without unexpected device-related adverse effects

DETAILED DESCRIPTION:
This is a research study to evaluate a new non-invasive drug-free acute treatment of headache in adolescents aged 12-17 years old. Participants are being asked to take part in this study because they suffer from persistent headaches.

Device description:

The device is a wireless wearable battery-operated stimulation unit controlled by a dedicated smartphone application. Treatments with Nerivio™ are self-administered by the user at the onset of a headache. The Nerivio™ includes several main components:

* A pair of electrodes covered with hydrogel and a removeable protective film
* An electronic circuitry and a battery
* A software that includes firmware and a software application for mobile platforms
* An armband to secure the attachment of the device and enable a discreet treatment

Procedures and duration of participation

Participants will receive a device and will be asked to treat headaches with it and report in the app the characteristics of the attacks at the beginning of the attack as well as at 2 hours after the treatment. The study includes 3 visits to the clinic. The investigators expect that participants will be in this research study for 8 weeks.

Why is this research study being done?

Participants are being asked to be in the study because they suffer from persistent headaches.

The Nerivio device is approved by the FDA for acute treatment of migraine with or without aura in patients 12 years of age or older. The purpose of this study is to assess the effect of the Nerivio device for treating New Daily persistent Headache (NDPH) in children. The Nerivio is a non-invasive device operated via a smartphone application that changes brain activity. The device is worn on the upper arm, and the treatment is self-administered at the headache onset. The device delivers non-painful electrical pulses to the skin that stimulate the body to initiate a pain inhibition mechanism in the brain. During the treatment, the users can adjust the intensity of the pulses according to how they tolerate it.

Marc DiSabella is the person responsible for this research study at Children's National. He is called the Principal Investigator.

What will happen in this research study?

Each participant will receive a device to be used at home for the acute treatment of their headaches. The device produces electrostimulation parameters aimed to relief headache pain. In addition, an app will be installed on the participants smartphone to control the device and record their headaches and their feedback regarding the effect of the device on their headaches.

Schedule of What the participants will do:

Enrollment Visit 1 (Day 0)

* Arrive to Children's National Medical Center with one of their parents, for their scheduled appointment. Bring packages of any medications that they are taking (for any medical condition).
* Eligibility assessment
* Meet with Dr. DiSabella or one of the colleagues and/or the study team to answer questions about their general health and their headaches.
* If this form is received today, the participant and their parent(s) can take time to read it carefully and make sure all of their questions and concerns are answered.
* The participant may request another appointment in case they would like to read this form at home and consult with family members or friends.
* If the participant is a girl and have had their first period, they will provide a urine sample for a pregnancy test.
* If the participant agree to participate, a member of the study staff will install the app on their smartphone. The investigators will provide an explanation on how to operate the smartphone application.
* the investigators will train the participant on how to complete their headache diary.

Run-in phase (Days 1-28)

* Complete the diary whenever the participant experience a new headache.
* The study staff will contact the participant to schedule their next visit

Device training Visit (Day 29-37)

* Eligibility to continue in the study will be assessed based on their reports and compliance in the run-in phase.
* The participant will receive a device.
* The investigator will train the participant how to use the device and find the intensity level that is best for them
* The participant can ask us any questions.
* The participant will take the Nerivio home with them.

Treatment phase Day 1-28 following visit 2

* Always have the device and their smartphone available.
* Use the device for the treatment of their headache onset (and always with 60 minutes of onset) and avoid taking rescue medication from the time of symptoms onset until 2 hours from treatment start (≈75 minutes from the end of the treatment). Report the 2-hour post treatment feedback through the smartphone application
* The application will ask the participant to rate their headache pain level at the beginning of the treatment, after 2 hours, and after 24 hours post treatment on a scale of 0-3 (0= no pain; 1= mild; 2= moderate; 3= severe)
* Call the study team if there is any change in their medical condition.
* At the end of this phase, the participant will be contacted by a member of the study team to schedule their next visit.

End of study visit 3. Please arrive to Children's National Medical Center for their scheduled appointment, complete the study questionnaires, if required and return the device.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age 12-17 years old at the time of informed consent, inclusive.
2. Participants have at least a 6-month history of headaches that meet the diagnostic criteria for New Daily Persistent Headache (NDPH)
3. Participants who are on stable dosing of prophylaxis agents for at least three months.
4. Participants have personal access to a smartphone (24/7)
5. Participants must be able and willing to comply with the protocol
6. Parents/Guardians must be able and willing to provide written informed consent
7. Participants must be able and willing to provide informed assent

Exclusion Criteria:

1. Participants with an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker, cochlear implant).
2. Participants with congestive heart failure (CHF), severe cardiac or cerebrovascular disease.
3. Participants with epilepsy.
4. Participants who have undergone nerve block (occipital or other) in the head or neck, or treatment with onabotulinum toxin A (Botox) to the head and/or neck in the prior four months.
5. Current participation in any other clinical interventional study
6. Participants without basic cognitive and motor skills required for operating a smartphone.
7. Pregnant or breastfeeding females
8. Participants who have previous experience with the device
9. Participants with arm circumference below 7.9 inches (20 cm)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Pain relief at 2 hours post-treatment | 2 hours post-treatment
  The proportion of participants achieving pain relief at 2 hours post-treatment in the test treatment, with no use of rescue/abortive medication (Pain relief defined as a change from severe to moderate, mild or none, moderate to mild or none, or mild to none)
Within-patient consistency | Before and at 1 Month after initiation of treatment with REN
  The repeatability of headache change, as described in the primary endpoint definition, in subsequent treated attacks. Thus, this endpoint measures the % of patient responding to the primary endpoint in at least 50% of their treated attacks
Disappearance of associated symptoms at 2 hours post-treatment | 2 hours post-treatment
  Disappearance of nausea, photophobia and phonophobia at 2 hours post- treatment
Functional disability at 2 hours post-treatment | 2 hours post-treatment
  The proportion of participants achieving a change of at least one grade in functional disability in the test treatment at 2 hours post-treatment with no use of rescue medication
Improve of quality of life assessed by PedsMIDAS questionnaire | Before and at 1 Month after initiation of treatment with REN
  Change in average headache disability as measured by PedsMIDAS before and at 1 month after initiation of treatment with REN.

CONTACTS AND LOCATIONS:
Overall Officials: Marc DiSabella, DO, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT05310227/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05310227/ICF_001.pdf